CLINICAL TRIAL: NCT04124159
Title: Risk of Recurrent Venous Thromboembolism in Patients With Provoked Deep Vein Thrombosis of the Leg and/or Pulmonary Embolism: a Prospective Cohort Study
Brief Title: Risk of Recurrent Venous Thromboembolism After Provoked Venous Thromboembolism
Acronym: AURECpro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sabine Eichinger, Principal investigator, Medical University of Vienna
Other Study IDs: AURECpro
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Recurrent Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous thromboembolism (VTE) is a common disease with an incidence of 1-2/1000 persons per year. VTE is a chronic disease with a considerable risk of recurrence. Patients with unprovoked VTE, i.e. VTE in the absence of a temporary risk factor including surgery, cancer or immobilisation, have a high recurrence risk and indefinite anticoagulation is generally recommended. The recurrence risk of patients with VTE provoked by a transient risk factor is regarded as low. Discontinuation of anticoagulation after three months is recommended because the benefit of reducing the recurrence risk further by prolonged anticoagulation is outweighed by the bleeding risk. However, the newer direct oral anticoagulants are potentially associated with a lower bleeding risk than vitamin K antagonists. Because they are also meanwhile widely available and are convenient there is a trend towards prolonging anticoagulation also in patients with a VTE after a transient provoking factor. However, the definition of transient provoking factors is imprecise and a distinct categorization according to the risk of recurrence is lacking. Preliminary evidence suggests that the recurrence risk varies considerably between the different transient provoking factors. In a prospective cohort study, the investigators will include patients with a deep vein thrombosis or pulmonary embolism provoked by a transient risk factor defined according to Guidance of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis (Kearon et al., J Thromb Haemost 2016; 14: 1480-3) after discontinuation of anticoagulation. The study endpoint is recurrent symptomatic VTE.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uni- or bilateral proximal or distal deep vein thrombosis of the leg and/or symptomatic pulmonary embolism provoked by a temporary risk factor
* Scheduled to be treated with anticoagulants for at least 3 months

Exclusion Criteria:

* Need for long-term anticoagulation
* Poor patient compliance
* No consent to participate
* VTE during pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive patients with a deep vein thrombosis and/or pulmonary embolism provoked by a transient risk factor after a minimum of 3 months of anticoagulation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
recurrent venous thromboembolism | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria